CLINICAL TRIAL: NCT04752709
Title: Clinical Study to Evaluate the Efficacy of Surface Electrical Stimulation for Urge Urinary Incontinence in Women
Brief Title: Efficacy of Surface Electrical Stimulation for Urge Urinary Incontinence in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elidah, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR-1155
Record Dates: First submitted 2021-01-22; First posted 2021-02-12 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-11

CONDITIONS: Urge Incontinence
Keywords: incontinence; bladder; urge; urgency; stimulation
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: Randomized between two active groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Device looks identical. A third person masks which software is coded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Group A (Experimental): Electrical muscle stimulator and surface applied electrode shaped to fit the perineal region, with stimulation group A.
  Interventions: Device: ELITONE UUI
- Active Group B (Active Comparator): Electrical muscle stimulator and surface applied electrode shaped to fit the perineal region with stimulation group B.
  Interventions: Device: ELITONE UUI

INTERVENTIONS:
Device: ELITONE UUI — External electrical stimulation
  Other Names: ELITONE muscle stimulator

SUMMARY:
The purpose of this research is to evaluate the effectiveness of the ELITONE-UUI electrical muscle stimulation device on treating urge incontinence. The aim of the device is to stimulate the pelvic floor muscles and surrounding structures to improve urinary incontinence.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate the effectiveness of the ELITONE-UUI electrical muscle stimulation device on treating urge incontinence in women. The aim of the device is to stimulate the pelvic floor muscles and surrounding structures to improve urinary incontinence. This is a randomized prospective controlled study of two active groups with a stimulation frequency difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Predominant urge urinary incontinence as determined by responses to a series of three standard questions from the King's Health Questionnaire; specifically:

  * An affirmative response to "Is it very difficult to control when you have a strong urge to urinate?",
  * An affirmative or negative response to "Do you lose urine with physical activities such as coughing, sneezing, running?",
  * And, if an affirmative response to the second question, an affirmative response to "Are more of your incontinence episodes due to a strong urge to urinate than to abdominal pressure such as sneezing?"
* Mild-moderate incontinence symptoms as determined by self-reported typical number of accidents of 1 or more per 24 hours. Symptom severity is later verified with data from the Daily Log (See 5.4)

Exclusion Criteria:

* Less than 1 incontinence accident (leak) per day*
* Severe incontinence as determined by self-reported >5 accidents per day
* Currently pregnant, may be pregnant, attempting to become pregnant, or delivery within previous 6 weeks
* Vaginal or pelvic surgery within previous 6 months
* Severe Obesity as defined by BMI >= 35
* Change in incontinence medication type or dosing within the last 3 months.
* History or symptoms of urinary retention, extra-urethral incontinence, overflow incontinence
* Pelvic pain/painful bladder syndrome
* Active urinary tract infection (UTI) or history of recurrent UTIs (more than three in a year), or recurrent vaginitis (bacterial/fungal)
* Tissues protruding outside the vagina at rest
* Presence of incontinence-associated dermatitis or other perineal skin disorders or lesions,
* Complete denervation of the pelvic floor
* Conductive inter-uterine devise (IUD/Coil) or metal implants in the abdominal or pelvic area, including the hip and lumbar spine,
* Chronic coughing
* Previous use of Interstim device or Botox for UI
* Implanted cardiac device, untreated cardiac arrhythmia or suffer from other heart problems.
* Cancer, epilepsy or cognitive dysfunction
* Underlying neurologic/neuromuscular disorder
* Impaired decision making, suicidal thoughts, or drug/alcohol dependence
* Lacks capacity to consent for themselves.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Kolb, M.S., Study Director — Elidah, Inc.
Locations (1):
- Elidah, Monroe, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Group A: Electrical muscle stimulator and surface applied electrode shaped to fit the perineal region, with stimulation group A (urge only for 6 seconds/cycle).
  ELITONE UUI: External electrical stimulation
- Active Group B: Electrical muscle stimulator and surface applied electrode shaped to fit the perineal region with stimulation group B (urge and stress)
  ELITONE UUI: External electrical stimulation
Period: Overall Study
Arm/Group | Active Group A | Active Group B
Started | 26 | 56
Completed | 17 | 34
Not Completed | 9 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Group A | Active Group B | Total
Number analyzed (Participants) | 17 | 34 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 23 | 36
  >=65 years | 4 | 11 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (13.8) | 57.8 (12.7) | 56.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 34 | 51
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 34 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Number of Urinary Incontinence Episodes Per Day
Description: The efficacy of a treatment for urinary incontinence measures how much the treatment changed urinary incontinence leakage from the beginning to the end of the 6 week period.
Time Frame: 6 weeks
Population: Total of 82 participants, but only 51 completed the trial.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Active Group A | Active Group B
Number analyzed (Participants) | 17 | 34
percentage change | 69.6 (30.9) | 66.1 (28.7)
Statistical Analysis 1: Comparison: Active Group A vs Active Group B; Test type: Other; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Safety Assessed by Number of Serious Adverse Events
Description: Any serious adverse events recorded during the trial.
Time Frame: 6 weeks
Population: There were no adverse events for any participants
Measure: Mean (Standard Deviation); unit: serious adverse events
Arm/Group | Active Group A | Active Group B
Number analyzed (Participants) | 17 | 34
serious adverse events | 0 (0) | 0 (0)

3. Secondary Outcome: Efficacy Assessed by Change in Incontinence Quality of Life Questionnaire (I-QOL)
Description: The efficacy assessed by change in Incontinence quality of life questionnaire (I-QOL). The scale is as follows: 1 = not at all , 2 = a little, 3 = moderately, 4 = quite a bit and 5 = extremely. The lower the value the less times it happens and the better outcome. A larger results indicate a higher change in I-QOL from beginning to end of trial. The minimum score total is 22 and maximum total score is 110.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: change of score on a scale
Arm/Group | Active Group A | Active Group B
Number analyzed (Participants) | 17 | 34
change of score on a scale | -26.6 (20.2) | -21.8 (15.9)

4. Secondary Outcome: Efficacy Assessed by Reduction in Average Pads Used Per Day
Description: Efficacy Assessed by Reduction in Average Pads used per day over the 6 week period.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Active Group A | Active Group B
Number analyzed (Participants) | 17 | 15
percentage of change | 27.8 (57.4) | 36.4 (33.5)

5. Secondary Outcome: Efficacy Assessed by Reduction in Average Bathroom Visits
Description: The efficacy assessed by average bathroom visits during the day and night.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Active Group A | Active Group B
Number analyzed (Participants) | 17 | 34
percentage of change | 5.9 (29.5) | 0.5 (26.0)

ADVERSE EVENTS:
Time Frame: 6 weeks of study
Arm/Group | Active Group A | Active Group B
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/34
Other Adverse Events (participants affected / at risk) | 0/17 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04752709/Prot_SAP_000.pdf